CLINICAL TRIAL: NCT02112513
Title: The Use of Maternal Serum Unconjugated Estriol for Monitoring the Prevention of Neonatal Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Haas, David M Haas, MD, MS, Indiana University
Other Study IDs: 1108006470
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Neonatal Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will obtain serum and saliva for estriol measurement before or within 2 hours of antenatal corticosteroid administration and about 24 hours after each dose is given.
  Women who consent to an optional PK portion of the study will have plasma samples obtained pre-dose and then on a schedule of approximately 0.5-2, 4-8, 10-15, 22-24 hours after the first dose and then 6-8, 24, and 48 hours after the 2nd dose. One sample will be collected in each of these times.
  A sample of whole blood will be obtained for DNA isolation. At the time of delivery, umbilical cord blood will be collected before being discarded for DNA and plasma. If we are unable to obtain umbilical cord blood, a buccal swab will be collected from the baby for DNA extraction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- salivary estriol measurement: Serum Estriol measurement via different assays is complex, expensive, labor intensive, time consuming, and generally performed at specific reference labs. Salivary Estriol level is an ideal potential surrogate for serum Estriol. It is convenient, non-invasive, and expedient. It may not, however, be as sensitive as serum estriol concentrations at detecting the association with glucocorticoid response. This study will collect both samples to determine which one is better suited for clinical use in this condition.
- serum estriol measure: we will determine if changes in maternal serum estriol represent a biomarker of response to antenatal corticosteroids as evidenced by neonatal development of RDS
- Betamethasone pharmacokinetic: we will determine if pharmacokinetic parameters and neonatal outcomes after antenatal corticosteroid use are associated with genetic polymorphisms in drug metabolizing enzymes, transporters, and steroid pathway genes
- betamethasone concentration and genetics: we will determine if maternal betamethasone concentrations and genetics are associated with maternal estriol changes or RDS development

SUMMARY:
The objective of this project is to evaluate clinical significance of measuring maternal blood estriol levels, after the administration of antenatal corticosteroids to enhance lung maturity. The investigators will test for associations of the change in maternal estriol with the development of respiratory distress syndrome. The investigators are also interested in determining whether salivary estriol is a valid surrogate to estriol blood assays. In addition the investigators will correlate these changes to pharmacokinetic (PK), pharmacodynamics (PD), and pharmacogenetic measures of betamethasone administration and fetal respiratory outcome

DETAILED DESCRIPTION:
We will obtain serum and saliva for estriol measurement before or within 2 hours of antenatal corticosteroid administration and about 24 hours after each dose is given.

Women who consent to an optional PK portion of the study will have plasma samples obtained pre-dose and then on a schedule of approximately 0.5-2, 4-8, 10-15, 22-24 hours after the first dose and then 6-8, 24, and 48 hours after the 2nd dose. One sample will be collected in each of these times.

A sample of whole blood will be obtained for DNA isolation. At the time of delivery, umbilical cord blood will be collected before being discarded for DNA and plasma. If we are unable to obtain umbilical cord blood, a buccal swab will be collected from the baby for DNA extraction.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 23-34 weeks with a diagnosis of threatened preterm labor or preterm premature rupture of membranes, or other diagnosis with a high likelihood of preterm delivery where the provider is recommending administering antenatal corticosteroids
* Singleton gestation
* Live fetus at the time of enrollment
* Being administered antenatal corticosteroids to enhance lung maturity
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* • Maternal age <18 years old

  * Major congenital anomalies
  * Multiple gestations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mothers with preterm labor (23 - 34 weeks) on antenatal corticosteroid for prevention of neonatal respiratory distress syndrome will be recruited
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11-08 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Respiratory distress syndrome | At least 30 days after delivery, the maternal and neonatal charts will be reviewed
  Respiratory Distress Syndrome is diagnosed clinically, by need for mechanical ventilation and oxygen for at least 48 hours, and the presence of radiologic chest findings.

CONTACTS AND LOCATIONS:
Overall Officials: David Haas, MD, MSc, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Will plan to deposit any genetic information into appropriate repository like dbgap. Other data potentially available upon request.
Supporting Information: Study Protocol
Time Frame: after study completion and will be available in dbgap as long as that database is supported
Access Criteria: contact study contact or dbgap